CLINICAL TRIAL: NCT01325922
Title: 50/50% Tilt and Tune Defibrillation Waveforms Utilizing High Voltage Lead Integrity Check Impedance
Brief Title: 50/50% Tilt and Tuned Defibrillation Waveform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Director, Clinical Affairs, St. Jude Medical
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: CRD 274
Record Dates: First submitted 2007-05-16; First posted 2011-03-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: DFT Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50/50% Tilt (Other)
  Interventions: Procedure: DFT Testing with a 50/50% tilt

INTERVENTIONS:
Procedure: DFT Testing with a 50/50% tilt

SUMMARY:
Study Description The purpose of this study is to compare the defibrillation efficacy between the 50/50% tilt biphasic waveform and the Tuned biphasic waveform utilizing High Voltage Lead Integrity Check (HVLIC) impedance.

Hypothesis The Tuned waveform reduces defibrillation thresholds (DFTs) when compared to the 50/50% tilt waveform.

Study Methods

* This is an acute, paired-sample, randomized (waveform testing sequence) study
* Patients are implanted with an Food and Drug Administration (FDA) approved St. Jude Medical (SJM) EpicTM+ DR/VR Implantable Cardioverter Defibrillator (or any other standard output ICD after Epic+) and defibrillation lead system.
* All study testing is completed at implant.
* Patients are randomized to begin DFT testing with either the 50/50% tilt or Tuned waveform.
* The HVLIC feature is used to measure the high voltage lead impedance and to program the Tuned and 50/50% tilt waveform pulse widths.
* The DFT is determined by an optimized binary search method that is designed to reduce the overall number of VF inductions to an average of 5.13 while maintaining very high resolution and accuracy.
* Total # of centers - 15 centers
* Sample size - 60 patients

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for ICD implantation.
* Patient is able to tolerate DFT testing.

Exclusion Criteria:

* Patient has a mechanical valve in the tricuspid position.
* Patient is pregnant.
* Patient is less than 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)